CLINICAL TRIAL: NCT05501080
Title: The Effect of Selective Adrenal Artery Embolization and Spironolactone on Ventricular Remodeling in Nondominant Lateral Secretory Primary Aldosteronism： A Randomized Controlled Clinical Study
Brief Title: The Effect of SAAE on Ventricular Remodeling in PA Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Yifei Dong, Professor, Second Affiliated Hospital of Nanchang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2022-073
Record Dates: First submitted 2022-08-12; First posted 2022-08-15 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Primary Aldosteronism
Keywords: primary aldosteronism; selective adrenal artery embolization; bilateral primary aldosteronism; Nondominant Lateral Secretory Primary Aldosteronism; Ventricular Remodeling
MeSH Terms: conditions — Hyperaldosteronism; Ventricular Remodeling | interventions — Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SAAE group (Experimental): Subjects received super selective adrenal artery embolization treatment
  Interventions: Other: Super selective adrenal artery embolization
- Spironolactone group (Active Comparator): Subjects received spironolactone treatment
  Interventions: Drug: Spironolactone

INTERVENTIONS:
Other: Super selective adrenal artery embolization — Superselective adrenal arterial embolization is an operation to inject embolic agent into adrenal artery through catheter to embolize part of adrenal gland, so as to reduce the secretion of adrenal hormone and reduce blood pressure.
  Arms: SAAE group
Drug: Spironolactone — Aldosterone receptor antagonists are recommended by guidelines for the treatment of bilateral primary aldosteronism.
  Arms: Spironolactone group

SUMMARY:
The study aims to assess the effect of superselective adrenal arterial embolization on ventricular remodeling in primary aldosteronism without lateralized aldosterone secretion by comparing it with spironolactone therapy.

DETAILED DESCRIPTION:
After being informed about the study and potential risks,all patients giving written informedconsent will undergo a 2-week screening period to determine eligibility for study entry.Atweek 0,patients who meet the eligibility requirements will be randomized in a 1:1 ratio to Superselective adrenal arterial embolization group or spironolactone therapy group.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age 18-60 years old, regardless of gender;
* (2) Blood pressure conditions meet one of the following: 1) Office blood pressure ≥ 140/90mmHg; 2) Ambulatory blood pressure monitoring whole day blood pressure > 130/80 mmHg or daytime blood pressure > 135/85 mmHg;
* (3) After strict drug elution, it met the diagnostic criteria of primary aldosteronism, and bilateral primary aldosteronism was confirmed by adrenal venous sampling;
* (4) No surgical intent or contraindication to surgery and willing to undergo pharmacological treatment or percutaneous superselective adrenal artery embolization;
* (5) The patient or his/her legal representative shall sign the written informed consent approved by the ethics committee before the screening.

Exclusion Criteria:

* (1) Primary hypertension or secondary hypertension with other causes;
* (2) A woman who is pregnant or lactating, or has a birth plan for the next year;
* (3) There are serious organic diseases, especially liver and kidney dysfunction(eGFR<45 mL/min/1.73 m2);
* (4) Severe allergy to contrast medium;
* (5) Other serious organic diseases, life expectancy < 12 months;
* (6) Adrenal CT showed adenoma.;
* (7) Patients are enrolled or want to participate in other clinical studies. During the enrollment study, the results of this study will be affected.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
LVMI | 12 months after SAAE
  Left ventricular mass index(LVMI)

SECONDARY OUTCOMES:
LVH | 12 months after SAAE
  left ventricular hypertrophy
ABPM | 1 month after SAAE
  24-hour ambulatory blood pressure monitor
ABPM | 12 months after SAAE
  24-hour ambulatory blood pressure monitor
PAC | 1 month after SAAE
  plasma aldosterone concentration
PAC | 12 months after SAAE
  plasma aldosterone concentration
PRA | 1 month after SAAE
  plasma renin activity
PRA | 12 months after SAAE
  plasma renin activity
ARR | 1 month after SAAE
  aldosterone-to-renin ratio
ARR | 12 months after SAAE
  aldosterone-to-renin ratio
Serum potassium | 1 month after SAAE
  Serum potassium
Serum potassium | 12 months after SAAE
  Serum potassium
serum creatinine | 1 month after SAAE
  serum creatinine
serum creatinine | 12 months after SAAE
  serum creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Yifei Dong, Doctorate, Study Director — Second Affiliated Hospital of Nanchang University
Locations (1):
- The Second Affiliated Hospital of Nanchang University, Nanchang, China

IPD SHARING:
Plan to Share IPD: No